CLINICAL TRIAL: NCT02769065
Title: A Phase 1 Safety, Tolerability, and Pharmacokinetic Study of Escalating Single and Multiple Oral Doses of TAK-071 in Healthy Subjects and Subjects With Mild Cognitive Impairment/Mild Alzheimer Disease and Relative Bioavailability and Food Effect of TAK-071 in Healthy Subjects
Brief Title: Study of TAK-071 in Healthy Participants and Participants With Mild Cognitive Impairment/Mild Alzheimer Disease and Relative Bioavailability (BA) and Food Effect of TAK-071 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated prematurely as data from cohort no longer needed due to indication change.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-071-1001; U1111-1176-7435 (Registry Identifier: WHO)
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer Disease; Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — TAK-071; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (30):
- SRD: Placebo Cohorts 1-6, 18 and 19 (Placebo Comparator): TAK-071 placebo-matching capsules, orally, once on Day 1 to non-Japanese healthy participants in the single-rising dose (SRD) period.
  Interventions: Drug: TAK-071 Placebo
- SRD: Cohort 1: TAK-071 1 mg (Experimental): TAK-071 1 mg, capsule, orally, once on Day 1 to non-Japanese healthy participants.
  Interventions: Drug: TAK-071
- SRD: Cohort 2: TAK-071 3 mg (Experimental): TAK-071 3 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on the 24-hour post-dose safety, tolerability and pharmacokinetic (PK) data from cohort 1.
  Interventions: Drug: TAK-071
- SRD: Cohort 3: TAK-071 9 mg (Experimental): TAK-071 9 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety, tolerability, and preliminary plasma PK and 12-hour CSF PK data.
  Interventions: Drug: TAK-071
- SRD: Cohort 4: TAK-071 20 mg (Experimental): TAK-071 20 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on the 24-hour post-dose safety and tolerability data from previous cohort.
  Interventions: Drug: TAK-071
- SRD: Cohort 5: TAK-071 40 mg (Experimental): TAK-071 40 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 will be based on 24-hour safety, tolerability, and preliminary plasma PK data from Cohort 4.
  Interventions: Drug: TAK-071
- SRD: Cohort 6: TAK-071 80 mg (Experimental): TAK-071 80 mg capsules, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety, tolerability, and preliminary plasma PK data from Cohort 5
  Interventions: Drug: TAK-071
- MRD: Placebo Cohorts 7-9 (Placebo Comparator): TAK-071 placebo-matching capsule, orally, once on Day 1 to non-Japanese healthy participants in the multiple-rising dose (MRD) period.
  Interventions: Drug: TAK-071 Placebo
- MRD: Cohort 7: TAK-071 3 mg (Experimental): TAK-071 3 mg capsules, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety and tolerability from Cohort 4 and the 24-hour preliminary plasma PK and 12-hour CSF PK data from Cohort 3.
  Interventions: Drug: TAK-071
- MRD: Cohort 8: TAK-071 9 mg (Experimental): TAK-071 9 mg capsules, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants. Dose of TAK-071 was based on safety, tolerability and available PK data arising from the ongoing SRD part and previous MRD cohort.
  Interventions: Drug: TAK-071
- MRD: Cohort 9: TAK-071 15 mg (Experimental): TAK-071 15 mg capsule, orally, once on Day 1, followed by a washout period of 7 days, then TAK-071 once daily for 21 days to non-Japanese healthy participants. Dose of TAK-071 will be based on safety, tolerability and available PK data arising from the ongoing SRD part and previous MRD cohort.
  Interventions: Drug: TAK-071
- MRD: TAK-071 Placebo Cohorts 10-12+Donepezil (Placebo Comparator): TAK-071 placebo-matching capsule, orally, once daily along with donepezil 5 mg, tablets, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants who were pre-treated with donepezil 5 mg, tablet, once daily for 3 weeks prior to administration of TAK-071.
  Interventions: Drug: Donepezil; Drug: TAK-071 Placebo
- MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg (Experimental): TAK-071 3 mg capsules, orally, once daily along with donepezil 5 mg, tablets, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants who were pre-treated with donepezil 5 mg, tablet, once daily for 3 weeks prior to administration of TAK-071. Dose of TAK-071 was same as the dose used in MRD Cohort 7.
  Interventions: Drug: TAK-071; Drug: Donepezil
- MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg (Experimental): TAK-071 9 mg capsules, orally, once daily along with donepezil 5 mg, tablets, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants who were pre-treated with donepezil 5 mg, tablet, once daily for 3 weeks prior to administration of TAK-071. Dose of TAK-071 was same as the dose used in MRD Cohort 8.
  Interventions: Drug: TAK-071; Drug: Donepezil
- MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg (Experimental): TAK-071 15 mg capsule, orally, once daily along with donepezil 5 mg, tablets, orally, once daily from Day 1 up to Day 21 to non-Japanese healthy participants who were pre-treated with donepezil 5 mg, tablet, once daily for 3 weeks prior to administration of TAK-071. Dose of TAK-071 was same as the dose used in MRD Cohort 9.
  Interventions: Drug: TAK-071; Drug: Donepezil
- MRD: Placebo Cohorts 13-15 (Experimental): TAK-071 placebo-matching capsule, orally, once on Day 1 to Japanese healthy participants.
  Interventions: Drug: TAK-071 Placebo
- MRD: Cohort 13: TAK-071 3 mg (Experimental): TAK-071 3 mg capsule, orally, once on Day 1, followed by a washout period of 7 days, then TAK-071 once daily for 21 days to Japanese healthy participants. Dose of TAK-071 was same as the dose used in MRD Cohort 7.
  Interventions: Drug: TAK-071
- MRD: Cohort 14: TAK-071 9 mg (Experimental): TAK-071 9 mg capsule or matching placebo, orally, once on Day 1, followed by a washout period of 7 days, then TAK-071 once daily for 21 days to Japanese healthy participants. Dose of TAK-071 was same as the dose used in MRD Cohort 8.
  Interventions: Drug: TAK-071
- MRD: Cohort 15: TAK-071 15 mg (Experimental): TAK-071 15 mg capsule, orally, once on Day 1, followed by a washout period of 7 days, then TAK-071 once daily for 21 days to Japanese healthy participants. Dose of TAK-071 was same as the dose used in MRD Cohort 9.
  Interventions: Drug: TAK-071
- Cohort 16 (Experimental)
  Interventions: Drug: TAK-071
- Bioavailability (BA)/Food Effect: Cohort 17 Sequence ABC (Experimental): A: TAK-071 10 mg capsule, orally once on Day 1 in the fasted state in Period 1, followed by B: TAK-071 10 mg tablet, orally, once on Day 1 in the fasted state in Period 2, followed by C: TAK-071 10 mg tablet, orally, once on Day 1 in the fed state in Period 3 in non-Japanese healthy participants. There was a 21-day washout after each period.
  Interventions: Drug: TAK-071
- BA/Food Effect: Cohort 17 Sequence BCA (Experimental): B: TAK-071 10 mg tablet, orally, once on Day 1 in the fasted state in Period 1, followed by C: TAK-071 10 mg tablet, orally, once on Day 1 in the Fed state in Period 2, followed by A: TAK-071 10 mg capsule, orally once on Day 1 in the fasted state Period 3 in non-Japanese healthy participants. There was a 21-day washout after each period.
  Interventions: Drug: TAK-071
- BA/Food Effect: Cohort 17 Sequence CAB (Experimental): C: TAK-071 10 mg tablet, orally, once on Day 1 in the fed state in Period 1, followed by A: TAK-071 10 mg capsule, orally once on Day 1 in the fasted state in Period 2, followed by B: TAK-20 10 mg tablet, orally, once on Day 1 in the fasted state in Period 3 in non-Japanese healthy participants. There was a 21-day washout after each period.
  Interventions: Drug: TAK-071
- SRD: Cohort 18: TAK-071 120 mg (Experimental): TAK-071 120 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety, tolerability, and preliminary plasma PK data from Cohort 6.
  Interventions: Drug: TAK-071
- SRD: Cohort 19: TAK-071 160 mg (Experimental): TAK-071 160 mg capsule, orally, once on Day 1 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety, tolerability, and preliminary plasma PK data from Cohort 18.
  Interventions: Drug: TAK-071
- SRD: TAK-071 Placebo+Donepezil Placebo (Placebo Comparator): TAK-071 placebo-matching capsule, orally, once on Day 1 followed by donepezil placebo-matching tablet, orally on Day 2 to non-Japanese healthy participants.
  Interventions: Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- SRD: TAK-071 Placebo+Donepezil (Placebo Comparator): TAK-071 placebo-matching capsule, orally, once on Day 1 followed by donepezil 10 mg tablet, orally, on Day 2 to non-Japanese healthy participants.
  Interventions: Drug: Donepezil; Drug: TAK-071 Placebo
- SRD: Cohort 20: TAK-071 40 mg+Donepezil (Experimental): TAK-071 40 mg capsule, orally, once on Day 1 followed by donepezil 10 mg, tablets, orally, once on Day 2 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety, tolerability, and preliminary plasma PK data from Cohort 19.
  Interventions: Drug: TAK-071; Drug: Donepezil
- SRD: Cohort 21: TAK-071 60 mg+Donepezil (Experimental): TAK-071 60 mg capsule, orally, once on Day 1 followed by donepezil 10 mg, tablets, orally, once on Day 2 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety and tolerability data from Cohort 20.
  Interventions: Drug: TAK-071; Drug: Donepezil
- SRD: Cohort 22: TAK-071 80 mg+Donepizil (Experimental): TAK-071 80 mg capsule, orally, once on Day 1, followed by donepezil 10 mg, tablets, orally, once on Day 2 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety and tolerability data from Cohort 21.
  Interventions: Drug: TAK-071; Drug: Donepezil

INTERVENTIONS:
Drug: TAK-071 — TAK-071 capsules
  Arms: BA/Food Effect: Cohort 17 Sequence BCA; BA/Food Effect: Cohort 17 Sequence CAB; Bioavailability (BA)/Food Effect: Cohort 17 Sequence ABC; Cohort 16; MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg; MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg; MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg; MRD: Cohort 13: TAK-071 3 mg; MRD: Cohort 14: TAK-071 9 mg; MRD: Cohort 15: TAK-071 15 mg; MRD: Cohort 7: TAK-071 3 mg; MRD: Cohort 8: TAK-071 9 mg; MRD: Cohort 9: TAK-071 15 mg; SRD: Cohort 18: TAK-071 120 mg; SRD: Cohort 19: TAK-071 160 mg; SRD: Cohort 1: TAK-071 1 mg; SRD: Cohort 20: TAK-071 40 mg+Donepezil; SRD: Cohort 21: TAK-071 60 mg+Donepezil; SRD: Cohort 22: TAK-071 80 mg+Donepizil; SRD: Cohort 2: TAK-071 3 mg; SRD: Cohort 3: TAK-071 9 mg; SRD: Cohort 4: TAK-071 20 mg; SRD: Cohort 5: TAK-071 40 mg; SRD: Cohort 6: TAK-071 80 mg
Drug: Donepezil — Donepezil over-encapsulated tablet
  Arms: MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg; MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg; MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg; MRD: TAK-071 Placebo Cohorts 10-12+Donepezil; SRD: Cohort 20: TAK-071 40 mg+Donepezil; SRD: Cohort 21: TAK-071 60 mg+Donepezil; SRD: Cohort 22: TAK-071 80 mg+Donepizil; SRD: TAK-071 Placebo+Donepezil
Drug: TAK-071 Placebo — TAK-071 placebo-matching capsules
  Arms: MRD: Placebo Cohorts 13-15; MRD: Placebo Cohorts 7-9; MRD: TAK-071 Placebo Cohorts 10-12+Donepezil; SRD: Placebo Cohorts 1-6, 18 and 19; SRD: TAK-071 Placebo+Donepezil; SRD: TAK-071 Placebo+Donepezil Placebo
Drug: Donepezil Placebo — Donepezil placebo-matching over-encapsulated tablet
  Arms: SRD: TAK-071 Placebo+Donepezil Placebo

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and pharmacokinetic (PK) of TAK-071 when administered as single rising dose (SRD) and multiple rising dose (MRD) orally in healthy participants and participants with mild cognitive impairment (MCI) or mild Alzheimer disease (AD).

DETAILED DESCRIPTION:
TAK-071 was being tested to find a safe and well-tolerated dose in healthy participants (non-Japanese and Japanese) and participants with MCI or mild AD (non-Japanese).

The study enrolled 179 participants. The study consisted of 4 parts: Single-rising dose (SRD) part (Cohorts 1-6, and 18-22), multiple-rising dose (MRD) part (Cohorts 7-15), Cohort 16 with 2-arm parallel design, and Cohort 17 relative bioavailability and food effect 3 period crossover design.

Participants in each cohort were randomized to receive treatment with TAK-071 or matching placebo using drug-in-capsule (DIC) in the morning following a minimum fast of 8 hours. In Cohort 16, participants were assigned to 1 of 2 possible treatments, TAK-071 or matching placebo. In Cohort 17, participants were assigned to 1 of 3 treatment sequences (ABC, BCA, or CAB) with treatment A being fasted state and capsule formulation, treatment B being fasted state and tablet formulation, and treatment C being fed state and tablet formulation. In Cohorts 20-22, participants were administered as a single dose of TAK-071 or placebo on Day 1, and a single dose of donepezil or placebo approximately 24 hours later on Day 2.

This multi-center trial was conducted in United States. The overall time to participate in this study was approximately 41 days. Participants made multiple visits to the clinic and were also contacted for the follow-up through the telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman who weighs at least 50 kg and has a body mass index (BMI) from 18.0 to 30.0 kg/m^2, inclusive, at Screening. Participants should be aged 18 to 55 years, inclusive (nonelderly at the time of informed consent and first study drug dose) for Cohorts 1 to 12, and 17 to 22; 20 to 55 years, inclusive, for Cohorts 13 to 15; and 55 to 90 years, inclusive, for participants in Cohort 16.
2. For Cohorts 13 to 15 only: First-generation Japanese, defined as having been born in Japan of Japanese parents and Japanese grandparents and living no more than 10 years outside of Japan, with no significant change in lifestyle, including diet, while living outside of Japan.
3. Cohort 16 only: Healthy elderly or participants with MCI or mild AD, who must have Mini Mental State Examination (MMSE) score of 18 to 30, inclusive or 18 to 26 inclusive, respectively, and no biomarker data to contradict this diagnosis. Participants with documented diagnosis of MCI or mild AD must be receiving ongoing donepezil therapy (10 mg) in the evening for a minimum of 21 days prior to Check-in (Day -1) or must consent to take donepezil dose titrated to at least 21 days of treatment with 10 mg QD prior to Check-in.

Exclusion Criteria:

1. Has clinically significant (Cohorts 1 to 15 and 17 to 22) or uncontrolled (Cohort 16) neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal (GI), urologic, immunologic, endocrine, or psychiatric disease or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. Has a history of type 1 diabetes (Cohorts 1 to 22) or type 2 diabetes (Cohorts 1 to 15, 17 to 22) or hemoglobin A1c >6.5% at Screening. Note: participants with controlled (hemoglobin A1c <7.0% at Screening) type 2 diabetes in Cohort 16 may participate in the study.
3. Has a risk of suicide or suicidal ideation with intent and plan according to the investigator's clinical judgment (affirmative answer to questions 4 and 5 of the ideation section of the Columbia-Suicide Severity Rating Scale) or has made a suicide attempt in the previous 6 months.
4. Cohort 16 only: Any significant neurologic disease (other than suspected incipient or mild AD), such as Parkinson disease, stroke, transient ischemic attack, multi-infarct dementia, Huntington disease, head trauma with clinically significant cognitive sequelae, or chronic central nervous system infection, per investigator discretion.
5. Has current or recent (within 6 months) GI disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United States from 05 May 2016 to 08 June 2017.
Pre-assignment Details: Healthy participants (non-Japanese and Japanese) and participants with mild cognitive impairment (MCI) or mild Alzheimer disease (AD) (non-Japanese) were enrolled in cohorts: TAK-071 single-rising-dose (SRD), multiple-rising dose (MRD), Food Effect Crossover or in combination with donepezil.
Groups:
- Cohort 16: TAK-071 capsule, orally, once on Day 1 for 21 days, followed by a washout period of 21 days, or placebo matching tablets, orally, once on Day 1 for 21 days. Donepezil was delivered as 5 mg tablet, orally, once followed by 10 mg tablet, orally, once in run-in period.
- SRD: Cohort 22: TAK-071 80 mg+Donepezil: TAK-071 80 mg capsule, orally, once on Day 1, followed by donepezil 10 mg, tablets, orally, once on Day 2 to non-Japanese healthy participants. Dose of TAK-071 was based on 24-hour safety and tolerability data from Cohort 21.
Period: Overall Study
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Cohort 16 | Bioavailability (BA)/Food Effect: Cohort 17 Sequence ABC | BA/Food Effect: Cohort 17 Sequence BCA | BA/Food Effect: Cohort 17 Sequence CAB | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Started | 17 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 0 | 4 | 4 | 4 | 6 | 6 | 9 | 9 | 5 | 6 | 6
Completed | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 0 | 4 | 4 | 4 | 6 | 6 | 9 | 9 | 5 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pre-treatment Event/Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who were enrolled and received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Cohort 16 | Bioavailability (BA)/Food Effect: Cohort 17 Sequence ABC | BA/Food Effect: Cohort 17 Sequence BCA | BA/Food Effect: Cohort 17 Sequence CAB | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 0 | 4 | 4 | 4 | 6 | 6 | 9 | 9 | 5 | 6 | 6 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (6.46) | 34.7 (4.32) | 32.8 (9.43) | 39.5 (11.33) | 41.7 (9.33) | 36.3 (8.16) | 29.7 (8.12) | 37.7 (6.56) | 33.2 (7.78) | 31.2 (8.59) | 39.2 (6.71) | 38.7 (6.31) | 36.5 (6.53) | 35.3 (7.17) | 36.7 (9.54) | 37.7 (3.79) | 38.2 (10.99) | 34.8 (6.42) | 36.2 (8.67) |  | 32.3 (7.37) | 38.3 (8.88) | 30.0 (2.45) | 31.8 (10.26) | 31.7 (6.95) | 38.0 (9.18) | 36.8 (9.82) | 38.6 (13.20) | 32.2 (6.77) | 35.8 (9.47) | 36.4 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 11
  Male | 15 | 4 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 |  | 4 | 4 | 4 | 6 | 6 | 7 | 8 | 4 | 6 | 4 | 166
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 1 | 2 | 2 | 3 | 1 | 0 | 2 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 |  | 0 | 1 | 1 | 2 | 1 | 5 | 2 | 1 | 1 | 3 | 41
  Not Hispanic or Latino | 14 | 3 | 6 | 5 | 4 | 4 | 3 | 5 | 6 | 4 | 3 | 5 | 4 | 6 | 4 | 3 | 5 | 5 | 5 |  | 4 | 3 | 3 | 4 | 5 | 4 | 7 | 4 | 5 | 3 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 5 | 5 |  | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 27
  Black or African American | 5 | 1 | 3 | 3 | 1 | 0 | 2 | 2 | 3 | 2 | 0 | 4 | 2 | 2 | 1 | 0 | 0 | 0 | 0 |  | 2 | 0 | 1 | 1 | 1 | 3 | 2 | 0 | 2 | 1 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  White | 8 | 3 | 2 | 3 | 4 | 5 | 3 | 4 | 2 | 4 | 5 | 1 | 4 | 3 | 4 | 0 | 0 | 0 | 0 |  | 1 | 4 | 3 | 5 | 3 | 6 | 6 | 3 | 3 | 5 | 94
  Multiracial | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 0 | 4 | 4 | 4 | 6 | 6 | 9 | 9 | 5 | 6 | 6 | 177
Height [Mean (Standard Deviation); unit: cm] | 175.8 (6.31) | 169.0 (5.97) | 175.0 (6.99) | 179.3 (8.14) | 172.3 (6.89) | 175.8 (7.31) | 179.8 (7.70) | 173.0 (9.63) | 178.8 (6.46) | 172.8 (5.12) | 174.7 (6.89) | 175.3 (6.53) | 177.0 (8.20) | 176.2 (4.54) | 168.0 (8.72) | 172.3 (2.08) | 171.2 (8.96) | 172.8 (6.10) | 178.2 (7.33) |  | 178.8 (5.06) | 175.8 (8.42) | 175.3 (5.80) | 173.0 (4.77) | 174.8 (5.56) | 175.2 (13.07) | 173.9 (7.61) | 178.4 (11.28) | 174.7 (5.47) | 170.8 (10.03) | 174.5 (9.64)
Weight [Mean (Standard Deviation); unit: kg] | 80.77 (7.563) | 71.80 (11.927) | 73.25 (12.314) | 85.35 (9.712) | 80.35 (7.076) | 82.58 (9.870) | 80.00 (10.942) | 78.05 (10.936) | 84.22 (11.284) | 76.73 (10.094) | 75.33 (14.062) | 81.93 (10.508) | 76.55 (8.147) | 76.23 (9.066) | 76.72 (9.972) | 69.63 (13.668) | 69.52 (7.253) | 67.72 (14.487) | 74.72 (12.583) |  | 79.73 (5.421) | 83.85 (11.356) | 75.53 (10.529) | 78.63 (12.980) | 78.42 (11.553) | 77.58 (12.727) | 77.66 (8.549) | 87.28 (11.637) | 72.25 (6.339) | 70.78 (10.039) | 77.09 (10.857)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 26.18 (2.349) | 24.99 (2.827) | 23.82 (3.090) | 26.50 (2.018) | 27.13 (2.766) | 26.65 (1.895) | 24.65 (1.895) | 26.04 (2.596) | 26.30 (2.966) | 25.71 (3.327) | 24.58 (3.503) | 26.59 (2.428) | 24.46 (2.344) | 24.52 (2.267) | 27.10 (2.066) | 23.38 (4.074) | 23.69 (1.113) | 22.56 (3.615) | 23.45 (3.032) |  | 24.95 (1.237) | 27.06 (2.221) | 24.66 (3.873) | 26.19 (3.611) | 25.60 (3.265) | 25.21 (2.721) | 25.66 (2.078) | 27.36 (1.767) | 23.73 (2.388) | 24.65 (1.432) | 25.30 (2.351)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 15 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 5 | 5 | 4 | 5 | 3 | 5 | 6 | 2 | 5 | 3 | 5 |  | 4 | 4 | 4 | 6 | 4 | 8 | 8 | 3 | 6 | 6 | 154
  Current Smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 0 |  | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 23
Alcohol Classification [Count of Participants; unit: Participants]
  Never Drunk | 12 | 5 | 6 | 6 | 6 | 4 | 6 | 6 | 5 | 6 | 4 | 5 | 6 | 3 | 5 | 2 | 4 | 5 | 4 |  | 4 | 4 | 3 | 6 | 4 | 8 | 8 | 5 | 6 | 6 | 154
  Current Drinker | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 1 |  | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 23
  Ex-drinker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xanthine/Caffeine Consumption [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 2 |  | 1 | 3 | 1 | 2 | 3 | 6 | 2 | 1 | 1 | 0 | 40
  No | 14 | 6 | 5 | 4 | 3 | 5 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 6 | 6 | 0 | 5 | 4 | 3 |  | 3 | 1 | 3 | 4 | 3 | 3 | 7 | 4 | 5 | 6 | 137
Female Reproductive Status [Count of Participants; unit: Participants]
  Postmenopausal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 6
  Surgically Sterile | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  Female of Childbearing Potential | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  N/A (Subject is Male) | 15 | 4 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 |  | 4 | 4 | 4 | 6 | 6 | 7 | 8 | 4 | 6 | 4 | 166

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs or gets worse after receiving study drug.
Time Frame: Day 1 up to Day 41
Population: Safety Analysis Set (SAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Bioavailability (BA)/Food Effect: Cohort 17 Regimen A: TAK-071 10 mg capsule, orally once on Day 1 in the fasted state in Period 1 or Period 2 or Period 3
- BA/Food Effect: Cohort 17 Regimen B: TAK-071 10 mg tablet, orally, once on Day 1 in the fasted state in Period 1 or Period 2 or Period 3
- BA/Food Effect: Cohort 17 Regimen C: TAK-071 10 mg tablet, orally, once on Day 1 in the fed state in Period 1 or Period 2 or Period 3
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 12 | 12 | 12 | 6 | 6 | 9 | 9 | 5 | 6 | 6
percentage of participants | 25.0 | 33.3 | 0 | 66.7 | 33.3 | 0 | 16.7 | 50.0 | 16.7 | 16.7 | 50.0 | 33.3 | 33.3 | 50.0 | 50.0 | 66.7 | 40.0 | 40.0 | 60.0 | 16.7 | 8.3 | 8.3 | 0 | 33.3 | 44.4 | 55.6 | 80.0 | 100 | 83.3

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Clinical Laboratory Tests at Least Once Post-dose
Description: Clinical laboratory tests included serum chemistry, hematology, coagulation and urinalysis. ULN=upper limit of normal range.
Time Frame: Day 1 up to Day 41
Population: SAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 12 | 12 | 12 | 6 | 6 | 9 | 9 | 5 | 6 | 6
percentage of participants
  Bilirubin (>2.0 mg/dL, >34.2 umol/L) | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase (>5*ULN) | 6.3 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (>30 mg/dL, >10.7 mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin Intl. Normalized Ratio (>1.5*ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (>3*ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post-dose
Description: Vital Sign measurements included systolic blood pressure (SBP), diastolic blood presssure (DBP), pulse, temperature, orthostatic SBP, orthostatic DBP and orthostatic pulse.
Time Frame: Day 1 up to Day 41
Population: SAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 12 | 12 | 12 | 6 | 6 | 9 | 9 | 5 | 6 | 6
percentage of participants
  Systolic Blood Pressure (SBP), Supine, <85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, Supine, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, 5 minutes (min) Supine, <85 mmHg, | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, 5 min Supine, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, 1 min Standing, <85 mmHg | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 20.0 | 8.3 | 8.3 | 0 | 16.7 | 0 | 0 | 11.1 | 0 | 0 | 0
  SBP, 1 min Standing, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, 3 min Standing, <85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 33.3 | 0 | 0 | 0 | 0 | 20.0 | 8.3 | 8.3 | 0 | 0 | 16.7 | 0 | 11.1 | 0 | 0 | 0
  SBP, 3 min Standing, >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (DBP), Supine, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, Supine, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, 5 min supine, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0
  DBP, 5 min Supine, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, 1 min Standing, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, 1 min Standing, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, 3 min Standing, <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0
  DBP, 3 min Standing, >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, Supine, <50 beats/min (bpm) | 6.3 | 33.3 | 0 | 0 | 0 | 16.7 | 16.7 | 16.7 | 0 | 16.7 | 0 | 0 | 33.3 | 50.0 | 50.0 | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, Supine, >120 beats/min | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, 5 min Supine, <50 beats/min | 25.0 | 0 | 16.7 | 0 | 33.3 | 16.7 | 16.7 | 33.3 | 0 | 33.3 | 0 | 16.7 | 33.3 | 16.7 | 16.7 | 33.3 | 60.0 | 40.0 | 20.0 | 33.3 | 41.7 | 25.0 | 66.7 | 0 | 44.4 | 22.2 | 40.0 | 33.3 | 16.7
  Pulse, 5 min Supine, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, 1 min Standing, <50 beats/min | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, 1 min Standing, >120 beats/min | 6.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 0 | 0 | 20.0 | 40.0 | 0 | 0 | 0 | 0 | 16.7 | 11.1 | 0 | 20.0 | 0 | 0
  Pulse, 3 min Standing, <50 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse, 3 min Standing, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 40.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0
  Temperature, <35.6 Celsius (C) | 0 | 0 | 16.7 | 0 | 0 | 0 | 33.3 | 50.0 | 16.7 | 33.3 | 16.7 | 16.7 | 33.3 | 0 | 33.3 | 66.7 | 40.0 | 20.0 | 60.0 | 25.0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 40.0 | 0 | 16.7
  Temperature, >37.7 C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Orthostatic SBP, 1 min Standing-Supine, <=-20 mmHg | 12.5 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 16.7 | 16.7 | 0 | 0 | 50.0 | 50.0 | 50.0 | 16.7 | 0 | 20.0 | 40.0 | 60.0 | 16.7 | 0 | 8.3 | 33.3 | 16.7 | 22.2 | 0 | 40.0 | 0 | 16.7
  Orthostatic SBP, 3 min Standing-Supine, <=-20 mmHg | 6.3 | 0 | 0 | 0 | 0 | 0 | 33.3 | 16.7 | 0 | 33.3 | 0 | 16.7 | 33.3 | 50.0 | 0 | 0 | 20.0 | 40.0 | 40.0 | 16.7 | 8.3 | 0 | 16.7 | 16.7 | 0 | 0 | 40.0 | 16.7 | 0
  Orthostatic DBP, 1 min Standing-Supine, <=-10 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 0 | 20.0 | 8.3 | 0 | 0 | 16.7 | 0 | 0 | 0 | 20.0 | 0 | 0
  Orthostatic DBP, 3 min Standing-Supine, <=-10 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 33.3 | 0 | 0 | 0 | 20.0 | 20.0 | 8.3 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0
  Orthostatic Pulse, 1 min Standing-Supine >10 bpm | 75.0 | 0 | 100 | 0 | 100 | 100 | 100 | 66.7 | 100 | 100 | 0 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 88.9 | 100 | 100 | 100 | 100
  Orthostatic Pulse, 3 min Standing-Supine >10 bpm | 75.0 | 0 | 100 | 0 | 100 | 100 | 100 | 66.7 | 100 | 100 | 0 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 88.9 | 100 | 100 | 100 | 100

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for 12-lead Electrocardiogram (ECG) Parameters at Least Once Post-dose
Description: A standard 12-lead electrocardiogram (ECG) was performed. The percentage of participants with markedly abnormal ECG findings during the study.
Time Frame: Day 1 up to Day 41
Population: SAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 5 | 5 | 12 | 12 | 12 | 6 | 6 | 9 | 9 | 5 | 6 | 6
percentage of participants
  ECG Mean Heart Rate (HR), <50 beats/min | 37.5 | 33.3 | 16.7 | 16.7 | 33.3 | 33.3 | 16.7 | 33.3 | 16.7 | 33.3 | 33.3 | 16.7 | 33.3 | 50.0 | 33.3 | 66.7 | 40.0 | 40.0 | 40.0 | 58.3 | 41.7 | 33.3 | 66.7 | 0 | 44.4 | 22.2 | 60.0 | 33.3 | 50.0
  ECG Mean HR, >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, Aggregate, <=80 millisecond (msec) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, Aggregate, >=200 msec | 18.8 | 0 | 16.7 | 0 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 16.7 | 16.7 | 16.7 | 66.7 | 0 | 40.0 | 20.0 | 33.3 | 25.0 | 25.0 | 0 | 0 | 11.1 | 11.1 | 20.0 | 0 | 16.7
  QRS Duration, Aggregate, <=80 msec | 31.3 | 33.3 | 33.3 | 0 | 50.0 | 16.7 | 16.7 | 33.3 | 16.7 | 16.7 | 16.7 | 50.0 | 16.7 | 16.7 | 16.7 | 33.3 | 40.0 | 20.0 | 40.0 | 8.3 | 16.7 | 16.7 | 16.7 | 50.0 | 11.1 | 11.1 | 20.0 | 0 | 16.7
  QRS Duration, Aggregate, >=180 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval, Aggregate, <=50 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval, Aggregate, >=460 msec | 12.5 | 33.3 | 16.7 | 0 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 20.0 | 20.0 | 16.7 | 16.7 | 8.3 | 16.7 | 0 | 11.1 | 11.1 | 40.0 | 0 | 0
  QTcB Interval, Aggregate, <=50 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB Interval, Aggregate ≥500 OR ≥30 and ≥450 msec | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 20.0 | 20.0 | 8.3 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0 | 0
  QTcF Interval, Aggregate, <=50 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval, Aggregate ≥500 OR ≥30 and ≥450 msec | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RR Interval, Aggregate, <=600 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 20.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RR Interval, Aggregate, >=1440 msec | 0 | 16.7 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 20.0 | 20.0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 11.1 | 11.1 | 0 | 0 | 0

5. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 Single-Rising Dose (SRD) Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine.
Measure: Median (Full Range); unit: hours
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.750 [1.48 to 4.00] | 4.017 [3.00 to 23.95] | 10.975 [3.00 to 24.00] | 8.000 [4.02 to 24.02] | 9.933 [3.00 to 48.00] | 24.033 [12.02 to 48.07] | 22.050 [8.00 to 39.95] | 24.058 [24.00 to 32.00]

6. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 Multiple-Rising Dose (MRD) Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: PK set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine.
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
hours | 2.500 [2.00 to 10.00] | 7.000 [3.00 to 12.00]

7. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
hours | 2.500 [2.00 to 6.00] | 4.000 [2.00 to 12.05]

8. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Full Range); unit: hours
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
hours | 24.058 [3.05 to 24.38]

9. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hour) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
hours | 11.017 [2.00 to 23.87]

10. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Mean (Full Range); unit: hours
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
hours | 3.000 [1.00 to 12.00]

11. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
hours | 4.000 [4.00 to 8.00] | 6.000 [2.00 to 12.00] | 12.000 [6.00 to 14.00]

12. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
hours | 4.000 [3.00 to 6.00] | 6.000 [6.00 to 23.75] | 8.000 [3.00 to 23.90]

13. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
hours | 4.000 [3.00 to 4.00] | 3.000 [1.50 to 6.05] | 3.000 [1.50 to 6.00]

14. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 3.508 [2.00 to 8.00] | 4.992 [3.00 to 10.00] | 7.000 [3.00 to 14.00]

15. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 3.500 [2.00 to 6.00] | 3.008 [2.00 to 4.00] | 3.500 [1.50 to 6.00]

16. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 21 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
hours | 4.983 [3.00 to 32.00] | 2.000 [1.00 to 8.00] | 6.000 [1.00 to 24.00]

17. Primary Outcome: Tmax: Time of First Occurrence of Cmax for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
hours | 26.000 [12.05 to 30.17] | 26.000 [4.02 to 27.00] | 30.000 [28.00 to 32.00]

18. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 Single-Rising Dose (SRD) Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 25.65 (5.8589) | 65.82 (5.4268) | 162.2 (36.548) | 328.0 (72.200) | 485.7 (240.47) | 901.7 (210.05) | 1292 (315.30) | 1387 (312.13)

19. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 Multiple-Rising Dose (MRD) Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
ng/mL | 74.33 (18.186) | 196.2 (54.668)

20. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
ng/mL | 244.5 (66.163) | 646.5 (95.032)

21. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
ng/mL | 264.8 (70.516)

22. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hour) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
ng/mL | 294.2 (57.007)

23. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 5
ng/mL | 936.4 (173.98)

24. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 78.98 (10.736) | 208.4 (47.773) | 278.0 (63.828)

25. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 81.16 (17.379) | 235.4 (37.740) | 329.6 (99.889)

26. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 235.6 (49.242) | 680.2 (181.99) | 895.2 (420.14)

27. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 79.12 (12.954) | 194.2 (17.325) | 303.7 (32.371)

28. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 232.8 (69.277) | 678.0 (67.620) | 970.7 (228.98)

29. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 1 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 219.7 (46.986) | 251.0 (41.946) | 242.5 (41.513)

30. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
ng/mL | 1110 (85.440) | 725.8 (186.03) | 532.2 (28.508)

31. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 Single-Rising Dose (SRD) Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 459.3 (111.88) | 1197 (92.810) | 3257 (634.89) | 6383 (1162.4) | 8905 (4529.9) | 16300 (3468.9) | 22350 (7203.2) | 25660 (8297.7)

32. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 Multiple-Rising Dose (MRD) Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
h*ng/mL | 1347 (302.98) | 3550 (765.01)

33. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg
Number analyzed (Participants) | 6 | 6
h*ng/mL | 4783 (1258.0) | 12520 (2132.7)

34. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
h*ng/mL | 5332 (1688.9)

35. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hour) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6
h*ng/mL | 5831 (998.50)

36. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 36 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 5
h*ng/mL | 19920 (4563.7)

37. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
h*ng/mL | 1485 (271.95) | 4201 (822.67) | 5581 (1141.6)

38. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Japanese Participants [Day 8]
Time Frame: Pre-dose on Day 8 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
h*ng/mL | 1529 (344.00) | 4634 (787.02) | 6110 (1217.2)

39. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Japanese Participants [Day 28]
Time Frame: Pre-dose on Day 28 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
h*ng/mL | 4439 (1135.6) | 13450 (3024.3) | 17120 (8088.8)

40. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 1]
Time Frame: Pre-dose on Day 1 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 1442 (251.62) | 3636 (286.83) | 5832 (921.06)

41. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 MRD Non-Japanese Participants [Day 21]
Time Frame: Pre-dose on Day 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 4467 (1461.6) | 13570 (1647.0) | 19210 (4669.4)

42. Primary Outcome: AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 21 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 16010 (4812.0) | 15190 (4576.6) | 16610 (5003.1)

43. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
h*ng/mL | 18370 (2361.9) | 12810 (2177.9) | 9440 (1353.7)

44. Primary Outcome: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points [up to 168 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1651 (644.79) | 5070 (3802.0) | 15640 (5944.7) | 30980 (5932.8) | 49550 (33766) | 106000 (19610) | 132700 (46773) | 162100 (69191)

45. Primary Outcome: AUC∞: Area Under the Concentration-Time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration for TAK-071 SRD Non-Japanese Participants TAK-071 + Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points [up to 168 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
h*ng/mL | 97640 (22123) | 48750 (12598) | 46370 (6094.8)

46. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1220 (397.35) | 3945 (1784.9) | 12450 (2466.5) | 26010 (3656.6) | 40240 (23644) | 90350 (13944) | 111700 (31926) | 133000 (45126)

47. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and multiple timepoints (up to 24 hrs) post-dose for Cohorts 7 and 8 and Pre-dose on Day 1 and multiple timepoints (up to 96 hrs) post-dose for Cohort 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 1347 (302.98) | 3550 (765.01) | 16880 (4514.9)

48. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 MRD Japanese Participants
Time Frame: Pre-dose on Day 1 and multiple time points (up to 96 hours) post-dose and Pre-dose on Day 8 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
h*ng/mL
  Day 1 | 3773 (968.76) | 11930 (2764.4) | 15790 (3273.2)
  Day 8 | 1529 (344.00) | 4634 (787.02) | 6110 (1217.2)

49. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 MRD Non-Japanese
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 1442 (251.62) | 3636 (286.83) | 5832 (921.06)

50. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 1 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 14210 (3392.5) | 13260 (2983.9) | 14610 (3324.3)

51. Secondary Outcome: AUClast: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
h*ng/mL | 85650 (13013) | 45970 (10798) | 41070 (4387.9)

52. Secondary Outcome: Terminal Disposition Phase Half-life (t1/2z) for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 50.894 [30.41 to 57.35] | 35.567 [23.34 to 132.30] | 54.998 [24.53 to 106.28] | 57.504 [41.58 to 84.66] | 53.219 [22.51 to 99.01] | 55.246 [32.94 to 68.05] | 51.933 [32.02 to 84.96] | 58.165 [32.58 to 87.60]

53. Secondary Outcome: Terminal Disposition Phase Half-life (t1/2z) for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 21 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
hours | 48.804 [23.44 to 92.82] | 50.590 [23.31 to 94.14] | 49.796 [23.35 to 100.82]

54. Secondary Outcome: Terminal Disposition Phase Half-life (t1/2z) for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
hours | 42.923 [40.47 to 67.70] | 33.505 [21.92 to 56.08] | 50.077 [37.37 to 63.32]

55. Secondary Outcome: CL/F: Apparent Clearance After Extravascular Administration for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 0.7222 (0.36130) | 0.7998 (0.36546) | 0.6494 (0.24348) | 0.6644 (0.12027) | 3.844 (7.3558) | 0.7762 (0.13868) | 1.008 (0.36826) | 1.141 (0.45838)

56. Secondary Outcome: CL/F: Apparent Clearance After Extravascular Administration for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 21 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
L/h | 0.6925 (0.27468) | 0.7232 (0.26191) | 0.6663 (0.25695)

57. Secondary Outcome: CL/F: Apparent Clearance After Extravascular Administration for TAK-071 SRD Non-Japanese Participants TAK-071+Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
L/h | 0.8453 (0.17228) | 1.304 (0.34484) | 0.8742 (0.11009)

58. Secondary Outcome: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L | 43.63 (10.532) | 44.96 (5.7176) | 48.10 (9.0985) | 54.62 (9.8917) | 321.0 (656.95) | 59.54 (11.499) | 70.25 (9.1042) | 84.47 (16.851)

59. Secondary Outcome: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for TAK-071 Relative Bioavailability and Food Effect
Time Frame: Pre-dose on Day 21 and multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C
Number analyzed (Participants) | 12 | 12 | 12
L | 44.43 (7.1688) | 46.74 (7.3595) | 43.82 (6.3235)

60. Secondary Outcome: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for TAK-071 SRD Non-Japanese Participants TAK-071 + Donepezil
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
Number analyzed (Participants) | 3 | 6 | 5
L | 59.03 (5.5208) | 62.40 (17.164) | 63.52 (11.895)

61. Secondary Outcome: Accumulation Ratio Based on AUCτ (Rac[AUC]) for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 21 and at multiple time points (up to 24 hours) post-dose for Cohorts 7 and 8 and Pre-dose on Day 28 and at multiple time points (up to 36 hours) post-dose for Cohort 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 5
Ratio | 3.568 (0.71765) | 3.713 (1.1916) | 3.778 (1.2626)

62. Secondary Outcome: Accumulation Ratio Based on AUCτ (Rac[AUC]) for TAK-071 MRD Japanese Participants
Time Frame: Pre-dose on Day 28 and at multiple time points [up to 24 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
Ratio | 2.973 (0.38747) | 3.241 (0.56613) | 3.096 (1.4212)

63. Secondary Outcome: Accumulation Ratio Based on AUCτ (Rac[AUC]) for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 21 and at multiple time points [up to 24 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 3.099 (0.75130) | 3.749 (0.55862) | 3.350 (0.92710)

64. Secondary Outcome: Accumulation Ratio Based on Plasma Cmax (Rac[Cmax]) for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 21 and at multiple time points [up to 24 hours] post-dose for Cohorts 7 and 8 and Pre-dose on Day 28 and at multiple time points (up to 36 hours) post-dose for Cohort 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 5
Ratio | 3.297 (0.59164) | 3.578 (1.2955) | 3.541 (0.86317)

65. Secondary Outcome: Accumulation Ratio Based on Plasma Cmax (Rac[Cmax]) for TAK-071 MRD Japanese Participants
Time Frame: Pre-dose on Day 28 and at multiple time points [up to 24 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
Ratio | 2.960 (0.26180) | 3.327 (0.74832) | 3.285 (1.5406)

66. Secondary Outcome: Accumulation Ratio Based on Plasma Cmax (Rac[Cmax]) for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 21 and at multiple time points [up to 24 hours] post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 2.929 (0.55096) | 3.527 (0.57233) | 3.257 (0.95527)

67. Secondary Outcome: AEt: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points [up to 96 hours] post-dose
Population: PK set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. Measurable TAK-071 was not detected in urine for Cohort 1 (TAK-071 1 mg). Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6
mg | 0.001731 (0.0015806) | 0.01632 (0.0062545) | 0.05753 (0.023868) | 0.08559 (0.052157) | 0.09052 (0.044805) | 0.1652 (0.097242) | 0.1505 (0.10905)

68. Secondary Outcome: AEt: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and 21 and at multiple time points (up to 24 hours) post-dose for Cohorts 7 and 8, and pre-dose on Day 1 and 28 and multiple time points (up to 96 hours) post-dose for Cohort 9
Population: PK set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. Here, number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 6
mg
  Day 1 | 0.001501 (0.0017987) | 0.005973 (0.0034636) | 0.04929 (0.019263)
  Day 21: number analyzed (Participants) | 6 | 6 | 0
  Day 21 | 0.009066 (0.0042349) | 0.02393 (0.014412) |
  Day 28: number analyzed (Participants) | 0 | 0 | 5
  Day 28 |  |  | 0.1119 (0.079021)

69. Secondary Outcome: AEt: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-071 MRD Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 96 hours) post-dose and pre-dose on Day 28 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
mg
  Day 1 | 0.003436 (0.0031125) | 0.02083 (0.0094853) | 0.03224 (0.023202)
  Day 28 | 0.01202 (0.010480) | 0.03394 (0.022682) | 0.06482 (0.062816)

70. Secondary Outcome: Fet: Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to Time t for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: fraction of drug excreted
Arm/Group | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6
fraction of drug excreted | 0.05771 (0.052687) | 0.1813 (0.069494) | 0.2877 (0.11934) | 0.2140 (0.13039) | 0.1131 (0.056006) | 0.1377 (0.081035) | 0.09408 (0.068159)

71. Secondary Outcome: Fet: Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to Time t for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Days 1 and 21 and at multiple time points (up to 24 hours) post-dose for Cohorts 7 and 8 and Pre-dose on Days 1 and 28 and multiple time points (up to 96 hours) post-dose for Cohort 9
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: fraction of drug excreted
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 6
fraction of drug excreted
  Day 1 | 0.05003 (0.059956) | 0.06636 (0.038484) | 0.3286 (0.12842)
  Day 21: number analyzed (Participants) | 6 | 6 | 0
  Day 21 | 0.3022 (0.14116) | 0.2659 (0.16013) |
  Day 28: number analyzed (Participants) | 0 | 0 | 5
  Day 28 |  |  | 0.7460 (0.52680)

72. Secondary Outcome: Fet: Fraction of Administered Dose of Drug Excreted in Urine From Time 0 to Time t for TAK-071 MRD Japanese Participants
Time Frame: as for outcome 69
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: fraction of drug excreted
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
fraction of drug excreted
  Day 1 | 0.1145 (0.10375) | 0.2314 (0.10539) | 0.2150 (0.15468)
  Day 28 | 0.4005 (0.34935) | 0.3771 (0.25202) | 0.4321 (0.41878)

73. Secondary Outcome: CLR: Renal Clearance for TAK-071 SRD Non-Japanese Participants
Time Frame: Pre-dose on Day 1 and at multiple time points [up to 96 hours] post-dose
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 6 | 6
L/h | 0.0006354 (0.00072647) | 0.001668 (0.00058267) | 0.002775 (0.00098052) | 0.002453 (0.0015795) | 0.001425 (0.00071797) | 0.001870 (0.0010016) | 0.001696 (0.0015594)

74. Secondary Outcome: CLR: Renal Clearance for TAK-071 MRD Non-Japanese Participants
Time Frame: Pre-dose on Days 1 and 21 and at multiple time points (up to 24 hours) post-dose for Cohorts 7 and 8 and Pre-dose on Days 1 and 28 multiple time points (up to 96 hours) post-dose for Cohort 9
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 6 | 6 | 6
L/h
  Day 1 | 0.001133 (0.0015553) | 0.001686 (0.00092928) | 0.003163 (0.0016448)
  Day 21: number analyzed (Participants) | 6 | 6 | 0
  Day 21 | 0.001937 (0.00099073) | 0.001991 (0.0012947) |
  Day 28: number analyzed (Participants) | 0 | 0 | 5
  Day 28 |  |  | 0.005431 (0.0032772)

75. Secondary Outcome: CLR: Renal Clearance for TAK-071 MRD Japanese Participants
Time Frame: as for outcome 69
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg
Number analyzed (Participants) | 5 | 5 | 5
L/h
  Day 1 | 0.0008641 (0.00063849) | 0.001783 (0.00090441) | 0.002093 (0.0016105)
  Day 28 | 0.002494 (0.0014594) | 0.002680 (0.0019001) | 0.003426 (0.0021244)

76. Secondary Outcome: CSF Cmax: Maximum Observed Concentration in Cerebrospinal Fluid (CSF) for TAK-071
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRD: Cohort 3: TAK-071 9 mg
Number analyzed (Participants) | 6
ng/mL | 0.008988 (0.0051582)

77. Secondary Outcome: CSF Cmax: Maximum Observed Concentration in Cerebrospinal Fluid (CSF) for TAK-071
Time Frame: Pre-dose on Day 28 and at multiple time points (up to 36 hours) post-dose
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 3
ng/mL | 0.01144 (0.0012682)

78. Secondary Outcome: CSF AUC(0-12): Area Under the CSF Concentration-time Curve From Time 0 to 12 Hours for TAK-071
Time Frame: Pre-dose on Day 1 and at multiple time points (up to 12 hours) post-dose
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SRD: Cohort 3: TAK-071 9 mg
Number analyzed (Participants) | 5
h*ng/mL | 13.68 (3.9324)

79. Secondary Outcome: CSF AUC(0-36): Area Under the CSF Concentration-time Curve From Time 0 to 36 Hours for TAK-071
Time Frame: Pre-dose on Day 28 and multiple time points (up to 36 hours) post-dose
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 3
h*ng/mL | 360.9 (73.780)

80. Secondary Outcome: Ratio of CSF AUC(0-12) to the Plasma AUC(0-12) for TAK-071
Time Frame: Pre-dose on Day 1 and at multiple time points [up to 168 hours] post-dose
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | SRD: Cohort 3: TAK-071 9 mg
Number analyzed (Participants) | 5
Ratio | 0.009098 (0.0034530)

81. Secondary Outcome: Ratio of CSF AUC(0-36) to the Plasma AUC(0-36) for TAK-071
Time Frame: Pre-dose on Day 28 and multiple time points (up to 36 hours) post-dose Cohort 9
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | MRD: Cohort 9: TAK-071 15 mg
Number analyzed (Participants) | 3
Ratio | 0.01140 (0.0014959)

82. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Donepezil MRD Non-Japanese Participants
Time Frame: Pre-dose on Days -1 and 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Day -1 | 3.000 [1.00 to 3.00] | 3.000 [2.00 to 4.00] | 3.008 [2.00 to 6.00]
  Day 21 | 2.508 [1.00 to 10.03] | 3.500 [2.00 to 8.00] | 2.500 [1.00 to 3.00]

83. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Donepezil MRD Non-Japanese Participants
Time Frame: Pre-dose on Days -1 and 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day -1 | 23.07 (3.6855) | 30.65 (5.9433) | 22.63 (4.2697)
  Day 21 | 26.58 (2.3659) | 29.95 (6.4071) | 25.97 (5.6163)

84. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post-dose for Donepezil
Time Frame: Pre-dose on Days -1 and 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  Day -1 | 410.1 (79.220) | 543.8 (113.62) | 399.5 (96.519)
  Day 21 | 472.5 (62.377) | 567.2 (135.33) | 430.5 (111.93)

85. Secondary Outcome: Ratio of Geometric Mean of Cmax for Donepezil After 21 Daily Doses of TAK-071
Description: A linear mixed effect model on the natural log-transformed parameters was performed with day as a fixed effect and participant as a random effect. Ratio is the exponentiated geometric mean value Day 21/Day -1 on the original scale.
Time Frame: Pre-dose on Days -1 and 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 68
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 8 | 8 | 8
Ratio | 1.160 [1.072 to 1.256] | 0.969 [0.914 to 1.028] | 1.121 [1.027 to 1.224]

86. Secondary Outcome: Ratio of Geometric Mean of AUC(0-24) for Donepezil After 21 Daily Doses of TAK-071
Description: as for outcome 85
Time Frame: Pre-dose on Days -1 and 21 and multiple time points (up to 24 hours) post-dose
Population: as for outcome 68
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg
Number analyzed (Participants) | 8 | 8 | 8
Ratio | 1.155 [1.059 to 1.260] | 1.055 [0.989 to 1.126] | 1.106 [1.014 to 1.207]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 41
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | SRD: Placebo Cohorts 1-6, 18 and 19 | SRD: Cohort 1: TAK-071 1 mg | SRD: Cohort 2: TAK-071 3 mg | SRD: Cohort 3: TAK-071 9 mg | SRD: Cohort 4: TAK-071 20 mg | SRD: Cohort 5: TAK-071 40 mg | SRD: Cohort 6: TAK-071 80 mg | MRD: Placebo Cohorts 7-9 | MRD: Cohort 7: TAK-071 3 mg | MRD: Cohort 8: TAK-071 9 mg | MRD: Cohort 9: TAK-071 15 mg | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg | MRD: Placebo Cohorts 13-15 | MRD: Cohort 13: TAK-071 3 mg | MRD: Cohort 14: TAK-071 9 mg | MRD: Cohort 15: TAK-071 15 mg | Cohort 16 | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A | BA/Food Effect: Cohort 17 Regimen B | BA/Food Effect: Cohort 17 Regimen C | SRD: Cohort 18: TAK-071 120 mg | SRD: Cohort 19: TAK-071 160 mg | SRD: TAK-071 Placebo+Donepezil Placebo | SRD: TAK-071 Placebo+Donepezil | SRD: Cohort 20: TAK-071 40 mg+Donepezil | SRD: Cohort 21: TAK-071 60 mg+Donepezil | SRD: Cohort 22: TAK-071 80 mg+Donepezil
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/5 | 0/5 | 0/5 | 0/0 | 0/12 | 0/12 | 0/12 | 0/6 | 0/6 | 0/9 | 0/9 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/5 | 0/5 | 0/5 | 0/0 | 0/12 | 0/12 | 0/12 | 0/6 | 0/6 | 0/9 | 0/9 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/16 | 2/6 | 0/6 | 4/6 | 2/6 | 0/6 | 1/6 | 3/6 | 1/6 | 1/6 | 3/6 | 2/6 | 2/6 | 3/6 | 3/6 | 2/3 | 2/5 | 2/5 | 3/5 | 0/0 | 2/12 | 1/12 | 1/12 | 0/6 | 2/6 | 4/9 | 5/9 | 4/5 | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRD: Placebo Cohorts 1-6, 18 and 19 (N=16) | SRD: Cohort 1: TAK-071 1 mg (N=6) | SRD: Cohort 2: TAK-071 3 mg (N=6) | SRD: Cohort 3: TAK-071 9 mg (N=6) | SRD: Cohort 4: TAK-071 20 mg (N=6) | SRD: Cohort 5: TAK-071 40 mg (N=6) | SRD: Cohort 6: TAK-071 80 mg (N=6) | MRD: Placebo Cohorts 7-9 (N=6) | MRD: Cohort 7: TAK-071 3 mg (N=6) | MRD: Cohort 8: TAK-071 9 mg (N=6) | MRD: Cohort 9: TAK-071 15 mg (N=6) | MRD: TAK-071 Placebo Cohorts 10-12+Donepezil (N=6) | MRD: Cohort 10: TAK-071 3 mg+Donepezil 5 mg (N=6) | MRD: Cohort 11: TAK-071 9 mg + Donepezil 5 mg (N=6) | MRD: Cohort 12: TAK-071 15 mg+Donepezil 5 mg (N=6) | MRD: Placebo Cohorts 13-15 (N=3) | MRD: Cohort 13: TAK-071 3 mg (N=5) | MRD: Cohort 14: TAK-071 9 mg (N=5) | MRD: Cohort 15: TAK-071 15 mg (N=5) | Cohort 16 (N=0) | Bioavailability (BA)/Food Effect: Cohort 17 Regimen A (N=12) | BA/Food Effect: Cohort 17 Regimen B (N=12) | BA/Food Effect: Cohort 17 Regimen C (N=12) | SRD: Cohort 18: TAK-071 120 mg (N=6) | SRD: Cohort 19: TAK-071 160 mg (N=6) | SRD: TAK-071 Placebo+Donepezil Placebo (N=9) | SRD: TAK-071 Placebo+Donepezil (N=9) | SRD: Cohort 20: TAK-071 40 mg+Donepezil (N=5) | SRD: Cohort 21: TAK-071 60 mg+Donepezil (N=6) | SRD: Cohort 22: TAK-071 80 mg+Donepezil (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 6 | 4
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02769065/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT02769065/SAP_001.pdf